CLINICAL TRIAL: NCT05176808
Title: Telehealth Parent-Implemented Intervention to Improve Social- Communication Outcomes in Young Children With ASD
Brief Title: Telehealth Parent-Implemented Intervention for Young Children With Autism Spectrum Disorder (ASD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00279093
Record Dates: First submitted 2021-12-08; First posted 2022-01-04 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Autistic Disorder; Active Autistic Disorder; Autism; Asperger Syndrome; PDD-NOS; Social Communication Delay; Mixed Expressive Receptive Language Disorder; Other Symbolic Dysfunctions
Keywords: Social Communication; Language; Engagement
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Communication; Language

STUDY DESIGN:
Intervention Model Description: Upon confirmation of eligibility and completion of the baseline assessments, participants will be randomly assigned to the TC or IPC study condition. Randomization will be done in randomly permuted groups of different sizes to reduce predictability of treatment assignment, with one half of the parent-child dyads in each block assigned to the IPC arm and one half assigned to the TC condition.
Who Masked: Outcomes Assessor
Masking Description: All participants will receive the same outcome battery of assessments. The individual evaluating the child and all coders will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Parent Coaching (TC) (Active Comparator): A family-centered, collaborative coaching approach, Practice-Based Coaching (Snyder et al., 2015), will be used. Coaches will use an NDBI coaching curriculum to support parents in targeting the child social-communication skills during interactions with their toddlers with ASD or social communication delays. The duration of the coaching period is 8-12 weeks with 2 sessions per week. Parents will be coached to implement NDBI strategies during daily routines with their young child with ASD or social communication delays following the coach and parent NDBI manuals developed in the primary principal investigator's lab. Trained study coaches will join families in their homes remotely via Kennedy Krieger Institute's secure Zoom password-protected account to provide coaching.
  Interventions: Behavioral: Early Achievements- Parent Coaching Intervention
- In-person Coaching(IPC) (Active Comparator): A family-centered, collaborative coaching approach, Practice-Based Coaching (Snyder et al., 2015), will be used. Coaches will use an NDBI coaching curriculum to support parents in targeting child social-communication skills during interactions with their toddlers with ASD or social communication delays. The duration of the coaching period is 8-12 weeks with sessions 2 times per week. Parents will be coached to implement NDBI strategies during daily routines with their young child with ASD following the coach and parent NDBI manuals developed in the primary principal investigator's lab. Coaching will be delivered in families' homes by trained study coaches to support parent implementation of NDBI strategies during daily life activities with their toddler with ASD or social communication delays.
  Interventions: Behavioral: Early Achievements- Parent Coaching Intervention

INTERVENTIONS:
Behavioral: Early Achievements- Parent Coaching Intervention — Children, along with a caregiver, will be randomized into one of two conditions to receive parent coaching guided by NDBI principles.

SUMMARY:
The primary objective of this research study is to improve outcomes involving core social-communication symptoms for young children with ASD or social communication delays by increasing access to clinically validated early behavioral intervention through a telehealth parent coaching model. The investigators will test the hypothesis that telehealth-delivered Naturalistic Developmental Behavioral Intervention parent coaching (TC) is non-inferior to in-person coaching (IPC) for the treatment of core social-communication symptoms in toddlers with either a social communication delay or ASD.

DETAILED DESCRIPTION:
The primary objective of this research study is to improve outcomes involving core social-communication symptoms for young children by increasing access to clinically validated early behavioral intervention through a telehealth parent coaching model. The investigators will test the hypothesis that telehealth-delivered Naturalistic Developmental Behavioral Intervention parent coaching (TC) is non-inferior to in-person coaching (IPC) for the treatment of core social-communication symptoms in toddlers with ASD. The secondary hypothesis is that feasibility (defined as parent fidelity) of TC is non-inferior to IPC. An exploratory objective is to guide clinical decision-making for telehealth implementation by examining the heterogeneity of treatment response across the two treatment arms. The investigators will test the hypothesis that baseline child behavioral dysregulation, active engagement, developmental quotient, and parent stress moderate child social-communication outcomes.

After completing eligibility testing, eligible children will be randomized into the TC or IPC condition. Each condition will involve twice weekly coaching sessions over 8-12 weeks. At the end of the intervention period, participants will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Meeting study criteria for ASD based on:

  * Autism Diagnostic Observation Schedule(ADOS) criteria for mild-to- moderate concern or greater (for children between 18 and 30 months) or algorithm cut-offs for ASD or autism (31-33 months),
  * Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)( criteria for ASD)
  * ASD diagnosis by clinician (clinical best estimate) by study team clinical research experts
* Meeting study criteria for social communication delay based on:

  * Scoring a T score of <35 on Expressive Language and/or Receptive Language subscales, Nonverbal developmental quotient of > 50 (Visual Reception and Fine Motor subscales averaged) AND Visual reception > 12 months
* Nonverbal developmental quotient (DQ) of > 63 based on the Visual Reception and Fine Motor subscales
* Gestational age of 36-42 weeks;
* Birth weight of > 2,500 grams;
* Absence of identifiable neurological (e.g., epilepsy), genetic (e.g., Down syndrome, fragile X, tuberose sclerosis, neurofibromatosis) or severe sensory- motor (e.g., cerebral palsy) conditions.
* Able to walk independently.
* Children must produce at least three different types of intentional directed (with eye contact or pairing vocalization and gesture) nonverbal or verbal communicative acts per day, with clear and specific examples, per parent report in the Eligibility Interview.

Exclusion Criteria:

* Having a primary language other than English
* Family lives >40 miles from a Kennedy Krieger Institute-Center for Autism Services, Sciences, and Innovation (CASSI) site.
* Child lives in foster care.

Ages: 18 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Child Duration of Joint Attention | 8-12 weeks
  10 minute caregiver/child play samples will be coded using an engagement coding schema. The schema differentiates different levels of engagement. This data will be used to compare duration of engagement states at pre- and post-testing.
Parent Fidelity of Implementation | 8-12 weeks
  Parent fidelity of implementation will be coded from the parent-child interaction sample obtained within the home at baseline and post-intervention by trained (to reliability) research assistants blind to group membership and timing of sample. This form consists of 26-items, where each item is rated using a 3-point Likert-type scale. Items reflect the key elements of Natural Developmental Behavioral Interventions (NDBI) which have been assessed in parent-implemented NDBI studies found to improve child social-communication outcomes. Ratings are based on effectiveness (well-timed, variety, developmental appropriateness) and frequency/consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.; Rachel Reetzke, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ingersoll B, Wainer AL, Berger NI, Pickard KE, Bonter N. Comparison of a Self-Directed and Therapist-Assisted Telehealth Parent-Mediated Intervention for Children with ASD: A Pilot RCT. J Autism Dev Disord. 2016 Jul;46(7):2275-84. doi: 10.1007/s10803-016-2755-z. PMID 26922192